CLINICAL TRIAL: NCT04380909
Title: Randomized Controlled Trial (RCT) to Evaluate the Efficacy of an Internet-based Self-help Program for People With Psychological Distress Due to Covid-19
Brief Title: ROCO - Self-help for People With Psychological Distress Due to the Covid-19 Situation
Acronym: ROCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-00990
Record Dates: First submitted 2020-05-07; First posted 2020-05-08 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Psychological Distress; Adjustment, Psychological; Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based self-help (Experimental): The self-help program consists of six text- and video-based modules. All participants in this group receive immediate access to the self-help program. The program's self-management approach does not provide for regular support from a specialist. However, participants can contact the study team if they need or want additional help.
  Interventions: Behavioral: Internet-based self-help
- Waiting control group (Other): Access to internet-based intervention after 3 weeks.
  Interventions: Behavioral: Internet-based self-help after 3 weeks

INTERVENTIONS:
Behavioral: Internet-based self-help — Six cognitive-behavioral, mindfulness and acceptance commitment based modules focusing on different aspects of psychological distress due to the Covid-19 situation.
  Arms: Internet-based self-help
Behavioral: Internet-based self-help after 3 weeks — Six cognitive-behavioral, mindfulness and acceptance commitment based modules focusing on different aspects of psychological distress due to the Covid-19 situation.
  Arms: Waiting control group

SUMMARY:
As part of the ROCO project, the University of Bern is investigating an online self-help program for people who are psychologically distressed due to the situation surrounding Covid-19. The ROCO program offers support in overcoming this psychological distress. ROCO stands for a 3-week online self-help program comprising 6 modules.

The aim of the study is to investigate the efficacy of an online self-help intervention for people with psychological distress due to the situation surrounding Covid-19. All participants will be randomized to one of two groups: The first group receives direct access to the online self-help intervention and the second group is a waiting control group that receives access to the program 3 weeks later. In both conditions additional care or treatment is allowed.

There are 4 assessments, which all take place online: baseline, post assessment (after 3 weeks) and two follow-up assessments (after 6 and 18 weeks). All participants from both groups are asked to fill out all assessments.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old
* Give a declaration of consent to participate in the study
* Have access to the internet
* Understand and master the German language to the degree that they understand the contents and instructions of the study
* Exceed a cut-off value of 4 points on the Brief Patient Health Questionnaire (PHQ-9; Löwe, Spitzer, Zipfel, & Herzog, 2002)
* Be able to specify an emergency address in the event of an acute crisis

Exclusion Criteria:

* Suicidal tendencies (SBQ-R Score ≥ 8)
* Existence of a known diagnosis of a psychotic or bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-07-29 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (Löwe et al., 2002) | up to 18 weeks
  9-item questionnaire assessing depressive symptoms

SECONDARY OUTCOMES:
Suicide Behavior Questionnaire Revised (Glaesmer et al., 2018) | up to 18 weeks
  4-item questionnaire assessing suicidal ideation
DASS-21: Depression, Angst, Stress-Skala (Lovibond & Lovibond, 1995) | up to 18 weeks
  21-item questionnaire assessing depression, anxiety and stress symptoms
SF-12: Short Form Health Survey (Ware et al., 1996) | up to 18 weeks
  12-item questionnaire assessing various aspects of well-being
LOT-R: Revised Life Orientation Test (Herzberg et al., 2006) | up to 18 weeks
  10-item questionnaire assessing optimism and pessimism
Berner Verbitterungsinventar Kurzversion (Znoj, 2008) | up to 18 weeks
  6-item questionnaire assessing embitterment
Emotion regulation skills SEK-27 (Berking & Znoj, 2008) | up to 18 weeks
  27-item questionnaire assessing emotion regulation skills
SWE: Skala zur Allgemeinen Selbstwirksamkeit (Jerusalem & Schwarzer, 2003) | up to 18 weeks
  10-item questionnaire assessing general self-efficacy
UCLA Loneliness Scale (Döring & Bortz, 1993) | up to 18 weeks
  9-item questionnaire assessing loneliness
Connor-Davidson Resilience Scale (Sarubin et al., 2015) | up to 18 weeks
  10-item questionnaire assessing resilience
ZUF-8: Zufriedenheitsfragebogen (Attkisson & Zwick, 1982) | at 3 weeks for experimental group and at 6 weeks for waiting control group
  8-item questionnaire assessing content with an online-program
SUS: System Usability Scale (Brooke, 1996) | at 3 weeks for experimental group and at 6 weeks for waiting control group
  10-item questionnaire assessing usability of an online-program

CONTACTS AND LOCATIONS:
Overall Officials: Hansjörg Znoj, Prof. Dr., Study Director — University of Bern; Thomas Berger, Prof. Dr., Principal Investigator — University of Bern
Locations (1):
- Universität Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brog NA, Hegy JK, Berger T, Znoj H. An internet-based self-help intervention for people with psychological distress due to COVID-19: study protocol for a randomized controlled trial. Trials. 2021 Mar 1;22(1):171. doi: 10.1186/s13063-021-05089-9. PMID 33648555